CLINICAL TRIAL: NCT07179159
Title: Efficacy and Safety of 14-Day Vonoprazan-Based Dual Therapy Versus Quadruple Therapy for Helicobacter Pylori Eradication: A Multicentre, Non-Inferiority Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yanqing Li (Other)
Collaborators: Longkou People's Hospital (Unknown); Qingdao Jimo People's Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Dezhou Hospital Qilu Hospital of Shandong University (Other); Zibo Maternal and Child Health Hospital (Unknown); Guanxian People's Hospital (Unknown); Yantai Zhifu Hospital (Unknown); The 2nd People's Hospital of Dongying City (Unknown); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Clinical Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202509
Record Dates: First submitted 2025-08-30; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: HELICOBACTER PYLORI INFECTIONS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 14-day vonoprazan-amoxicillin dual therapy (Experimental)
  Interventions: Drug: 14-day vonoprazan-amoxicillin dual therapy
- 14-day vonoprazan-amoxicillin-levofloxacin-bismuth quadruple therapy (Active Comparator)
  Interventions: Drug: 14-day vonoprazan-amoxicillin-levofloxacin-bismuth quadruple therapy
- 14-day vonoprazan-amoxicillin-clarithromycin-bismuth quadruple therapy (Active Comparator)
  Interventions: Drug: 14-day vonoprazan-amoxicillin-clarithromycin-bismuth quadruple therapy

INTERVENTIONS:
Drug: 14-day vonoprazan-amoxicillin dual therapy — vonoprazan 20mg bid + amoxicillin 1000mg bid
  Arms: 14-day vonoprazan-amoxicillin dual therapy
Drug: 14-day vonoprazan-amoxicillin-levofloxacin-bismuth quadruple therapy — vonoprazan 20mg bid + amoxicillin 1000mg bid + levofloxacin 500mg qd + bismuth 220mg bid
  Arms: 14-day vonoprazan-amoxicillin-levofloxacin-bismuth quadruple therapy
Drug: 14-day vonoprazan-amoxicillin-clarithromycin-bismuth quadruple therapy — vonoprazan 20mg bid + amoxicillin 1000mg bid + clarithromycin 500mg bid + bismuth 220mg bid
  Arms: 14-day vonoprazan-amoxicillin-clarithromycin-bismuth quadruple therapy

SUMMARY:
This study is a multicentre, non-inferiority randomized controlled trial to compare the efficacy and safety of 14-day vonoprazan-based dual therapy with versus quadruple therapy for the eradication of Helicobacter pylori. The primary outcome is eradication rate, and the secondary outcome includes the incidence of adverse events and compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years, male or female
2. Current Helicobacter pylori infection (positive 13C-urea breath test)
3. No prior Helicobacter pylori eradication therapy

Exclusion Criteria:

1. Severe underlying conditions, such as hepatic insufficiency, renal insufficiency, malignant tumours
2. Active gastrointestinal bleeding
3. History of upper gastrointestinal surgery
4. History of drug hypersensitivity
5. Use of bismuth compounds or antibiotics within the past 4 weeks, or acid-suppressing agents within the past 2 weeks
6. Pregnant or lactating women
7. Presence of other risk-increasing behaviours such as alcohol abuse or illicit drug use
8. Individuals unable or unwilling to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
eradication rate | 6 weeks after treatment

SECONDARY OUTCOMES:
adverse events | immediately after a 2-week treatment
compliance | immediately after a 2-week treatment
  Satisfactory compliance was defined as taking medications with at least 80% of the prescribed dosage. The proportion of patients with satisfactory compliance was calculated among all patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China